CLINICAL TRIAL: NCT06895889
Title: A Prospective, Randomized, Controlled, Open-label, First-in-human Phase I/IIb Study to Evaluate the Safety and Efficacy of the EB-OC Graft in the Repair of Full Thickness Chondral/osteochondral Defects of the Knee
Brief Title: EB-OC for the Treatment of Focal Chondral/Osteochondral Defects in the Knee
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Epibone, Inc. (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EB-OC-01
Record Dates: First submitted 2025-02-06; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Chondral Defect; Osteochondral Defect
Keywords: Abrasion Chondroplasty; Focal Chondra; Osteochondral Defects; Orthobiologics; Cartilage regeneration

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 2:1 ratio to the investigational product or control, with participants randomized to control provided the crossover opportunity for EB-OC graft treatment at 12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- EB-OC graft (Experimental): This group will receive the EB-OC graft via an arthrotomy procedure. An arthrotomy is an open joint procedure.
  Interventions: Device: EB-OC Graft Implantation
- Abrasion Chondroplasty (Active Comparator): This group will receive abrasion chondroplasty. Abrasion chondroplasty is a minimally invasive procedure.
  Interventions: Procedure: Abrasion chondroplasty

INTERVENTIONS:
Device: EB-OC Graft Implantation — The implantation of the EB-OC graft is completed via an arthrotomy, which is categorized as a minor surgery and is done on an outpatient basis, which means you can go home the same day. It is completed under general anesthesia and may last between one to two hours.
  Arms: EB-OC graft
Procedure: Abrasion chondroplasty — Abrasion chondroplasty is a minimally invasive procedure in which the surgeon uses a rotary burr to scrape off the bone tissue from the surface of the joint.
  Arms: Abrasion Chondroplasty

SUMMARY:
EB-OC is a tissue engineered osteochondral tissue graft comprising of a living tissue engineered cartilage layer attaching to a bone scaffold. The goal of this clinical trial is to learn about in the safety and efficacy of the EB-OC graft in participants who require repair of chondral/osteochondral defects of the knee. The main question it aims to answer is if the EB-OC graft works to regenerate osteochondral tissue comprising of native hyaline cartilage anchors to the regenerated bone. Participants will receive treatment of either the EB-OC Graft implantation in an arthrotomy procedure or abrasion chondroplasty. Researchers will compare results from the EB-OC graft to abrasion chondroplasty to assess overall safety and effectiveness.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, open-label, first-in-human Phase I/IIb study to evaluate the safety and efficacy of the EB-OC graft in the repair of full thickness chondral/ osteochondral defects of the knee as compared to abrasion chondroplasty. Enrollment in this study is expected to occur over 12 months. Subjects will be evaluated for safety and efficacy for 24 months post-surgery. It is anticipated that the study will be completed in approximately 36 months.

EB-OC comprising of a living tissue engineered cartilage layer attaching to a bone scaffold. The living tissue engineered cartilage layer is a cartilage-like tissue grown in the lab from an allogeneic (from donor) bone-marrow derived mesenchymal stem cells that have been induced to under cartilage development refered as Drug Substance EB-CMB.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female, between 18 and 65 years of age
2. Subject's body mass index (BMI) is ≤ 35 kg/m2.
3. Subject has up to two symptomatic, full-thickness cartilage defects of the knee femoral condyle with or without bone involvement that are:

   1. Located on the femoral condyles or femoral trochlea
   2. Each between 0.75 and 3 cm2 in area on screening images as confirmed by an independent radiologist
   3. Classified as International Cartilage Repair Society (ICRS) grade 3 or 4.
   4. Has baseline Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain <65 and KOOS Activities of Daily Life <70.
4. Subject is willing and able to provide informed consent and comply with study requirements.
5. Subject agrees to actively participate in a strict rehabilitation protocol and follow-up program.
6. For women of childbearing potential, subject must have a negative pregnancy test at Screening, cannot be lactating and must be willing to use adequate contraception throughout study participation.

   Note: Adequate contraception methods will include the following: Abstinence, Oral Contraceptives, Barrier Methods (Condoms, IUD's), or surgical sterilization.
7. Subject is willing to give up the use of narcotics for 6 months post-surgery and use and record alternative pain medications (e.g., acetaminophen, or narcotic analgesics, if prescribed).

Note: Post-surgical use of aspirin for clot prevention and narcotics for immediate post-surgical pain are acceptable.

Exclusion Criteria:

1. Lesions on the opposing surface of the tibia that are classified as ICRS grade 3 or 4.
2. Lesions on the opposing surface of the patella that are classified as ICRS grade 3 or 4 if a trochlear defect is being treated.
3. Any existing prosthetic implants in the index knee.
4. History of knee surgery in the index knee within 6 months prior to screening.
5. Has osteoarthritis of Kellgren-Lawrence Grade ≥3 as diagnosed on standing radiographs in the index knee.
6. Known history of hypersensitivity to gentamicin, other aminoglycosides, or products of bovine origin.
7. Inflammatory arthritis, inflammatory joint disease, or uncorrected congenital blood coagulation disorders.
8. Current infection or history of infection in the index knee joint.
9. Current skin infection of the index knee joint or skin infection of the index knee joint within the past 3 months.
10. Osteochondral defect greater than 7 mm in depth.
11. Avascular necrosis (AVN) or osteonecrosis (ON).
12. Meniscus tears or defects that require concomitant or prior removal of >50% of meniscus in the index knee.
13. Varus or valgus malalignment exceeding 5° in either knee.
14. Need for corrective concomitant osteotomy (tibio-femoral or patellofemoral).
15. Symptomatic musculoskeletal condition in the lower limbs that could impede efficacy measures in the target knee.
16. Diagnosed musculoskeletal cancer or any diagnosed cancer, other than musculoskeletal if not on long term remission (e.g., at least 5 years or negative biopsy at last exam), except basal cell carcinoma.
17. Clinically significant abnormalities in vital signs at the time of screening defined by

    * Systolic BP >140 or <90 mmHg or diastolic BP >90 or <60 mmHg
    * Pulse <60 or >100 bpm
    * Respiratory Rate <9 or >20
    * Temperature >99 °F
18. Hemoglobin, platelet, white blood cell count, creatinine, aspartate aminotransferase (AST), and alanine aminotransferase (ALT), prothrombin time (PT), and partial thromboplastin time (PTT) below the lower limit of normal or above the upper limit of normal.
19. Active infection (e.g., HIV, viral hepatitis, syphilis, cellulitis, respiratory infection, etc.).
20. Alcohol and drug (including medication) abuse.
21. Subjects with any contraindications to MR imaging.
22. Participation in concurrent trials or in previous trial within 90 days of signing informed consent.

Intra-Operative Exclusion Criteria

1. Greater than 2 defects requiring treatment
2. A symptomatic defect with greater than 5 mm of bone loss

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of adverse event incidents as compared to control | 12 months
  Number of adverse event incidents based on clinical laboratory and vital signs during the 12-month period post-surgery as compared to control
Adverse event incident rate (% pateint) as compared to control | 12 months
  Adverse event incident rate (% patient) based on clinical laboratory and vital signs during the 12-month period post-surgery as compared to control
Number of adverse events based on electrocardiogram readout as compared to control | Day 1, 1 week post Surgery
  Number of adverse events based on Electrocardiogram (ECG) readout as compared to control
Incident rate of adverse event (% patient) based on electrocardiogram readout as compared to control | Day 1, 1 week post Surgery
  Incident rate of adverse event (% patient) based on Electrocardiogram (ECG) readout as compared to control
Report of all adverse events including incidence, timing, severity, and relationship to the treatment | 36 months
  The incidence, timing, severity, and relationship to treatment of all Adverse Events (AE), will be collected and coded using Medical Dictionary for Regulatory Activities (MedDRA).
Report of secondary surgical interventions | 36 months
  Any secondary surgical interventions required to treat the target defects (e.g., reoperations, supplemental fixation, or other interventions) will be recorded.

SECONDARY OUTCOMES:
Patient reported outcome KOOS scores | 5 weeks, 3 months, 6 months, 12 months, 18 months, and 24 months
  KOOS scores which assesses Pain, Symptoms, Activities of Daily Living, Sport and Recreation Function, and Quality of Life. Score of 0-100 with zero being worst and 100 being best outcome
Patient reported outcome IKDC scores | 5 weeks, 3 months, 6 months, 12 months, 18 months, and 24 months
  IKDC Score (Subjective Knee Evaluation, Evaluator Global Assessment and Patient Global Assessment). Score of 0-100 with zero being worst and 100 being best outcome
MRI AMADEUS score | Screening, 12 months
  MRI AMADEUS score of the treated defect at Screening. Score 0-100 with 0 represents worst case cartilage defect and 100 represents best intact cartilage and bone
MRI MOCART score | 12 months
  MRI MOCART scoring of the treated defect. Score ranging from 0-100 with 0 being worst and 100 being best.
Descriptive report of graft integration based on clinical evaluation | 12 months
  Descriptive clinical evaluation of graft integration based on CT image.

CONTACTS AND LOCATIONS:
Overall Officials: Sarindr Bhumiratana, PhD, Study Director — Epibone, Inc.